CLINICAL TRIAL: NCT02574390
Title: Answer ALS -Creation of a Large Bio-repository of iPS Cells, Cell Lines, and Bio-fluid Samples, Combined With Clinical Information to Rapidly Advance Therapeutics That Could Treat ALS
Brief Title: Answer ALS: Individualized Initiative for ALS Discovery
Acronym: AnswerALS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Massachusetts General Hospital (Other); Emory University (Other); Ohio State University (Other); Washington University School of Medicine (Other); Cedars-Sinai Medical Center (Other); University of California, Irvine (Other); Massachusetts Institute of Technology (Other); New York Genome Center (Other); Leandro P. Rizzuto Foundation (Other); Texas Neurology (Unknown); Northwestern University Les Turner ALS Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00082277
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Flail Arm ALS; Progressive Muscular Atrophy; Monomelic Amyotrophy; Motor Neuron Disease; Asymptomatic ALS Gene Carriers; Healthy Controls
Keywords: ALS; stem cell; biomarker; disease progression
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Muscular Atrophy, Spinal; Amyotrophy, monomelic; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — plasma, serum, DNA, Cerebrospinal fluid, induced pluripotent stem cells,
Oversight: Data Monitoring Committee: No

SUMMARY:
Creation of a large repository of induced pluripotent stem cells (iPSC), bio-fluid samples (blood and spinal fluid (optional)), and cell lines for ALS gene identification. This will be combined carefully with collected measures of the pattern of the symptoms people with ALS have and how these change over time. People with other motor neuron diseases and healthy controls will be included as comparisons

DETAILED DESCRIPTION:
Patients will have 5 study visits; screening, 3, 6, 9 and 12 months. There will be a one year post-participation follow-up period, during which they will receive an email or phone call interview once every 3 months. During the first year, samples will be collected, breathing, muscle strength, spasticity, general function and cognitive behavior will be assessed. Healthy controls will have 2 study visits during which blood samples will be collected and questionnaires given.

ELIGIBILITY:
Inclusion Criteria:

* Participants with familial or sporadic ALS diagnosed as possible, laboratory-supported probable, probable or definite according to the World Federation of Neurology (WFN) El Escorial criteria, Primary Lateral Sclerosis Flail Arm ALS, Progressive Muscular Atrophy, Monomelic Amyotrophy, Motor Neuron Disease, Asymptomatic ALS Gene Carriers
* Participants who are ages 18-100, inclusive.

Exclusion Criteria:

* Participants with Spinal-Bulbar Muscular Atrophy
* Known diagnosis of HIV/AIDS, Hepatitis B, or Hepatitis C.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with ALS, Primary Lateral Sclerosis Flail Arm ALS Progressive Muscular Atrophy Monomelic Amyotrophy Motor Neuron Disease Asymptomatic ALS Gene Carriers
Sampling Method: Non-Probability Sample
Enrollment: 1049 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) | once every 3 months for one year
  12 questions about patient's ability to function in certain activities of daily living. Each question is out of 4 with 4 being normal and 0 being completely impaired.
ALS Cognitive Behavioral Scale (ALS-CBS) | once every 3 months for one year
  short measure of cognition and behavior in patients with ALS. The cognitive portion consists of 8 tasks with a perfect score being 20. The behavioral portion measures changes in personality and behavior since the onset of ALS symptoms as well as mood, pseudobulbar affect and fatigue and is completed by a family member or caregiver. A normal score is 45.
Slow Vital Capacity (SVC) | once every 3 months for one year
  measurement of the maximum amount of air that can be exhaled following a deep breath.
Strength Testing with Hand Held Dynamometer (HHD) | once every 3 months for one year
  muscle strength testing performed on upper and lower limbs, ankles, wrists and fingers using a small hand held device. These measurements are followed over time and compared to measure decline.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Maragakis, MD, Principal Investigator — Johns Hopkins University; James D Berry, MD, Principal Investigator — Massachusetts Generel Hospital
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Texas Neurology, Dallas, Texas